CLINICAL TRIAL: NCT07164248
Title: Retrospective Evaluation of Bone Mineral Density Measurements, Clinical Indications, and Risk Factors for Osteopenia/Osteoporosis in Female Adolescents Attending at a Tertiary Care Center
Brief Title: Evaluation of Bone Mineral Density Indications and Outcomes in Female Adolescents: Implications for Early Detection of Osteopenia/Osteoporosis and Gynecologic Practice
Acronym: TEEN-BMD
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nursen Kurtoglu Aksoy, Obstetrics and Gynecology Specialist, Bagcilar Training and Research Hospital, Bagcilar Training and Research Hospital
Other Study IDs: 2025/05/05/048
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Bone Density; Osteopenia; Amenorrhea; Primary Amenorrhea
Keywords: Osteoporosis; Amenorrhea; DEXA; Adolescent; Bone Health; Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic; Amenorrhea; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 - Adolescent gynecology referrals: Patients referred for DEXA scans due to gynecologic indications such as hypogonadism, amenorrhea, premature ovarian insufficiency [POI], functional hypothalamic amenorrhea [FHA], or hypogonadotropic hypogonadism
- Cohort 2 - Referrals from other specialties: Patients referred for DEXA scans by other departments, such as pediatrics, endocrinology, or additional medical specialties

SUMMARY:
This retrospective study evaluates bone mineral density (BMD) measurements obtained by dual-energy X-ray absorptiometry (DEXA) in adolescent girls aged 12 to 21 years at a tertiary care center. The study focuses on patients referred from the adolescent gynecology clinic as well as from other medical specialties.

Key objectives are:

Comparing the BMD indications and results requested from the gynecology department with the indications and BMD results requested from other departments. Thus, the BMD scores of patients with hypogonadism can be compared with other groups at risk for bone health.

To assess BMD Z-scores across specific gynecologic diagnoses, including premature ovarian insufficiency, functional hypothalamic amenorrhea (FHA), and hypogonadotropic hypogonadism.

To analyze the relationship between gynecologic clinical features-such as age at menarche and duration of amenorrhea-and BMD Z-scores.

By combining clinical, hormonal, and densitometric data, this study aims to identify risk factors for low bone density in adolescents, support earlier recognition of osteopenia/osteoporosis, and provide guidance for appropriate interventions in adolescent gynecology practice.

DETAILED DESCRIPTION:
Adolescence is a critical period for bone mass acquisition, and disturbances during this stage may predispose to osteopenia or osteoporosis in later life. Various clinical conditions encountered in gynecology, endocrinology, and other specialties may require evaluation of bone mineral density (BMD). However, data on referral indications and bone health outcomes in adolescents remain scarce.

This retrospective study focuses on female adolescents aged 12-21 years who underwent dual-energy X-ray absorptiometry (DEXA) scans at a tertiary care center. The cohort includes patients referred from the adolescent gynecology clinic as well as those referred from other medical departments.

The study objectives are:

To compare referral indications for BMD testing between gynecology and other specialties.

To evaluate differences in BMD Z-scores across specific gynecologic diagnoses, including premature ovarian insufficiency (POI), functional hypothalamic amenorrhea (FHA), and hypogonadotropic hypogonadism.

To examine the relationship between clinical features (such as age at menarche and duration of amenorrhea) and BMD outcomes within the gynecology group.

The analysis will provide insight into how referral patterns, gynecologic and endocrine conditions, and clinical characteristics influence bone health in adolescent girls. By highlighting risk factors for low BMD, the study aims to support earlier recognition and management of bone health problems in this population.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescents aged 12-21 years
* Underwent bone mineral density (BMD) measurement with DEXA at the study center between 2020 and 2025
* Available clinical and biochemical records, including referral indication

Exclusion Criteria:

* Incomplete or missing BMD scan data
* Insufficient clinical information in medical records
* Patients with underlying conditions unrelated to bone health that preclude accurate evaluation (e.g., major skeletal deformities interfering with DEXA interpretation)

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Female adolescents aged 12-21 years who underwent bone mineral density (BMD) measurement by dual-energy X-ray absorptiometry (DEXA) at a tertiary care hospital. The study includes patients referred from the adolescent gynecology clinic as well as those referred from other medical specialties (e.g., pediatrics, endocrinology).
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) Z-scores in Adolescent Girls | At the time of DEXA scan (retrospective chart review, 2020-2025
  Comparison of BMD Z-scores between adolescents (12-21 years) referred from the adolescent gynecology clinic and those referred from other specialties.

CONTACTS AND LOCATIONS:
Overall Officials: Nursen Kurtoglu, Principal Investigator — Bagcilar Training and Research Hospital
Locations (1):
- Bagcilar Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. The study is retrospective and based on medical records, and patient confidentiality restrictions prevent data sharing.